CLINICAL TRIAL: NCT05962177
Title: Montpellier PROspective Cohort in Relapsing Remitting Multiple Sclerosis Using Imaging and Serologic
Acronym: PROMISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL20_0422
Record Dates: First submitted 2023-06-15; First posted 2023-07-27 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; MRI; Longitudinal cohort; Real life; Biomarkers
MeSH Terms: conditions — Multiple Sclerosis | interventions — Magnetic Resonance Spectroscopy; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Relapsing-remitting Multiple sclerosis benefiting from a moderately effective treatment (Experimental): Moderately effective treatment includes interferon beta, glatiramer acetate, Teriflunomide, dimethyl Fumarate and monomethyl fumarate n= 175 patients
  Interventions: Other: Magnetic Resonance Imaging; Other: Blood withdrawal; Other: Neuropsychological tests
- Relapsing-remitting Multiple sclerosis benefiting from a highly effective treatment (Experimental): Highly effective treatment includes Natalizumab, Ocrelizumab, Rituximab, Ofatumumab, Fingolimod and Cladribine n= 175 patients
  Interventions: Other: Magnetic Resonance Imaging; Other: Blood withdrawal; Other: Neuropsychological tests
- Untreated relapsing-remitting Multiple sclerosis (Experimental): Patients untreated for relapsing-remitting Multiple sclerosis n= 50 patients
  Interventions: Other: Magnetic Resonance Imaging; Other: Blood withdrawal; Other: Neuropsychological tests

INTERVENTIONS:
Other: Magnetic Resonance Imaging — Magnetic Resonance Imaging
Other: Blood withdrawal — Blood withdrawal
Other: Neuropsychological tests — Neuropsychological tests

SUMMARY:
Several prospective monocentric cohorts of between 250 and 1000 patients have been set up in order to characterize more precisely the evolution of the disease. Nevertheless, due to an initial recruitment carried out in the years 2000-2010, they do not constitute a faithful representation of the patients followed in clinical routine, in particular in terms of distribution of treatments. Indeed, the introduction, about 10 years ago, of high efficacy treatments (HET) has changed the management of the disease and a significant proportion of patients not controlled by medium efficacy treatments (MET) of the disease are now stable on HET. Nevertheless, if their short-term efficacy has been clearly demonstrated, it remains important to be able to confirm the superiority of HET over MET with the help of prospective cohorts (thus ensuring a retention of patients > 90% over the long term) analyzing all clinical and imaging biomarkers, imaging and biological data.

The measurement of cerebral atrophy and its progression is probably one of the most interesting and most easily used biomarkers that can be used clinically to assess this silent progression in these groups of patients.

The progression of brain atrophy is also dependent on many other non-modifiable but also modifiable factors outside of MS that need to be better evaluated and eventually managed.

Nevertheless, the existence of various neurological comorbidities (sleep disorders, headaches) on this atrophy has not been specifically analyzed to date. The functional assessments used in routine follow-up are most often performed in a care facility and have many limitations: lack of reproducibility, inter/intra operator variability, poor correlation with functional and quality of life scales, etc.

It is therefore extremely important to be able to identify new clinical biomarkers of disease progression of the disease by evaluating the physical capacities of the patients as precisely as possible.

This study is a single-center, prospective cohort study of a population of 400 patients with relapsing remitting MS (RRMS).

The main objective of this study is to compare, on morphological imaging criteria (T1 volumetry), the progression of brain atrophy (biomarker of disease progression) at 3 years in RRMS patients according to treatment line (MET vs HET).

DETAILED DESCRIPTION:
Several prospective monocentric cohorts of between 250 and 1000 patients have been set up in order to characterize more precisely the evolution of the disease. Nevertheless, due to an initial recruitment carried out in the years 2000-2010, they do not constitute a faithful representation of the patients followed in clinical routine, in particular in terms of distribution of treatments. Indeed, the introduction, about 10 years ago, of high efficacy treatments (HET : Natalizumab, Fingolimod, Ocrelizumab, Rituximab, Ofatumumab, Cladribine) has changed the management of the disease and a significant proportion of patients not controlled by medium efficacy treatments (MET : Beta interferons, glatiramer acetate, teriflunomide, dimethyl fumarate, monomethyl fumarate) of the disease are now stable on HET. Nevertheless, if their short-term efficacy has been clearly demonstrated, it remains important to be able to confirm the superiority of HET over MET with the help of prospective cohorts (thus ensuring a retention of patients > 90% over the long term) analyzing all clinical and imaging biomarkers, imaging and biological data.

The measurement of cerebral atrophy and its progression is probably one of the most interesting and most easily used biomarkers that can be used clinically to assess this silent progression in these groups of patients.

The progression of brain atrophy is also dependent on many other non-modifiable but also modifiable factors outside of MS that need to be better evaluated and eventually managed.

Nevertheless, the existence of various neurological comorbidities (sleep disorders, headaches) on this atrophy has not been specifically analyzed to date. The functional assessments used in routine follow-up are most often performed in a care facility and have many limitations: lack of reproducibility, inter/intra operator variability, poor correlation with functional and quality of life scales, etc.

It is therefore extremely important to be able to identify new clinical biomarkers of disease progression of the disease by evaluating the physical capacities of the patients as precisely as possible.

This study is a single-center, prospective cohort study of a population of 400 patients with relapsing remitting MS (RRMS).

The main objective of this study is to compare, on morphological imaging criteria (T1 volumetry), the progression of brain atrophy (biomarker of disease progression) at 3 years in RRMS patients according to treatment line (MET vs HET).

3 groups of interest will be studied and included in the study:

* Group 1: RRMS with medium efficacy treatment (interferon beta, glatiramer acetate, Teriflunomide, dimethyl fumarate, monomethyl fumarate) of the disease (n=175 patients)
* Group 2: RRMS with high efficacy treatment (Natalizumab, Ocrelizumab, Rituximab, Ofatumumab, Fingolimod, Cladribine: n=175 patients)
* Group 3: Untreated RRMS (n=50 patients)

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 and under 60 years of age
* Patients with Relapsing-remitting MS without relapse for at least 6 months
* EDSS<6 at time of inclusion

Exclusion Criteria:

* Secondary progressive MS or Primary progressive MS at time of inclusion
* Evidence of disease progression (clinical or radiological)
* Change in treatment within 6 months prior to inclusion
* Subject with a contraindication to MRI (claustrophobia, pacemaker, etc.)
* Inability to follow the follow-up planned by the study
* Pregnant or breastfeeding women
* Patient not affiliated to the social security system or not benefiting from such a system
* Adult protected by law or patient under guardianship or curatorship
* Failure to obtain written informed consent after a reflection period

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Total brain atrophy | 3 years after Day 1
  Total brain atrophy measured with T1 MRI scans

SECONDARY OUTCOMES:
Quantitative analysis: analysis of FLAIR hypersignals number | 3 years after Day 1
  Analysis of FLAIR hypersignals numbers (lesion load)
Quantitative analysis: analysis of FLAIR hypersignals volume | 3 years after Day 1
  Analysis of FLAIR hypersignals volume
Qualitative analysis: analysis of central vein lesions | 3 years after Day 1
  Identification and quantification of central vein lesions on SWI
Qualitative analysis: analysis of peripheral rim lesion | 3 years after Day 1
  Identification and quantification of peripheral rim lesions on SWI
Quantitative analysis: measurement of mean diffusivity | 3 years after Day 1
  measurement of the mean diffusivity using diffusion tensor analysis
Quantitative analysis: measurement of anisotropy fraction | 3 years after Day 1
  measurement of anisotropy fraction using diffusion tensor analysis
Quantitative analysis: measurement of cerebral blood flow (CBF) | 3 years after Day 1
  cerebral blood flow analysis on 3DPCASL
Changes in serum light chain neurofilament values | 3 years after Day 1
  Changes in serum light chain neurofilament values in patients with RRMS patients according to the treatment line (high efficacy treatment vs. medium efficacy treatment)
Clinical assessment scale: relapses | 3 years after Day 1
  Clinical assessment scales (absolute changes and reaching threshold values): Relapses
Clinical assessment scale: Expanded Disability Status Scale (EDSS) | 3 years after Day 1
  The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist.
Clinical assessment scale: Computerized Speed Cognitive Test (CSCT) | 3 years after Day 1
  " Computerized Speed Cognitive Test " (CSCT) provides screening for cognitive impairment in MS patients
Clinical assessment scale: Six-Minute Walk Test (6MWT) | 3 years after Day 1
  Six-Minute Walk Test
Clinical assessment scale: 9-Hole Peg Test (9-HPT) | 3 years after Day 1
  The 9-HPT is a brief, standardized, quantitative test of upper extremity function.
Clinical assessment scale: Timed 25-Foot Walk (T25-FW) | 3 years after Day 1
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk.
Quality of life scale: The 5-level EQ-5D questionnaire (EQ5D-5L) | 3 years after Day 1
  EQ5D5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Lower score indicate better outcomes.
  The questionnaire also includes a visual analog scale in which the patient quantifies his or her perception of quality of life using a score ranging from the worst imaginable state of health (0) to the best imaginable state of health (100).
Quality of life scale: The Brief Pain Inventory (BPI) | 3 years after Day 1
  The Brief Pain Inventory (BPI) assesses the severity of pain and its impact on functioning.
Quality of life scale: DN4 | 3 years after Day 1
  The "Douleur Neuropathique 4 questions" questionnaire is a 4 questions questionnaire on neuropathic pain rating from 0 to 10; If the patient's score is 4/10 or more, the test is positive When the practitioner suspects neuropathic pain, the DN4 questionnaire is useful as a diagnostic tool.
Fatigue scale: Chalder Fatigue Scale | 3 years after Day 1
  Chalder Fatigue Scale is a self-administered questionnaire for measuring the extent and severity of fatigue.
Fatigue scale: Modified Fatigue Impact Scale (MFIS) | 3 years after Day 1
  Modified Fatigue Impact Scale (MFIS) provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning.
Sleep scale: Epworth Sleepiness Scale (ESS) | 3 years after Day 1
  The Epworth Sleepiness Scale (ESS) is used to assess daytime sleepiness.The ESS is a self-administered questionnaire with 8 questions. ESS score can range from 0 to 24. A global score greater than ten is diagnostic of excessive daytime sleepiness .
Depression scale: Beck Depression Inventory (BID) | 3 years after Day 1
  The Beck Depression Inventory (BDI) contains 21 items and identifies symptoms and attitudes associated with depression.
Anxiety scale: Generalized Anxiety Disorder 7-Item Scale (GAD-7) | 3 years after Day 1
  Generalized Anxiety Disorder 7-Item Scale measures seven anxiety symptoms.
Headaches scale: ef-ID Migraine | 3 years after Day 1
  ef-ID Migraine guide towards the diagnosis of migraine
Exploratory criteria:Serum Glial Fibrillary Acidic Protein (GFAP) | 3 years after Day 1
  Serum GFAP
Exploratory criteria: Pittsburgh Sleep Quality Index (PSQI) questionnaire | 3 years after Day 1
  Evaluation of habitual sleep quality trough a validated questionnaire. 19 items where each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Exploratory criteria: Idiopathic Hypersomnia Severity Hypersomnia Scale (IHSS) | 3 years after Day 1
  Patient-reported questionnaire assessing the severity of excessive sleepiness, prolonged sleep duration, cognitive impairment and sleep inertia. The total score ranges from 0 to 50, with higher scores indicating more severe symptoms.
Exploratory criteria: RU SATED score | 3 years after Day 1
  The Regularity, Sleep Quality, Alertness, Timing, Efficiency, Duration scale for sleep (RU SATED) ranges from 0 to 30, with higher scores indicating better sleep health.
Exploratory criteria: Insomnia Severity Index (ISI) | 3 years after Day 1
  The Insomnia Severity Index is a seven item-scale scored on a five-point scale (from 0 to 4). The total score ranges from 0 to 28. Higher scores indicate more insomnia.
Exploratory criteria: Headaches Impact Test (HIT-6) | 3 years after Day 1
  HIT-6 addresses six main domains affected by headaches, including pain, social functioning, role functioning, cognitive functioning, vitality and psychological stress.
  Little or no impact: 49 or less ; some impact: 50-55 ; substantial impact: 56-59 ; severe impact: 60-78
Exploratory criteria: Godin Leisure-Time Exercise Questionnaire (GLTEQ) | 3 years after Day 1
  Godin Leisure-Time Exercise Questionnaire (GLTEQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Neurology Department, Hopital Gui de Chauliac, Montpellier, France

IPD SHARING:
Plan to Share IPD: No